CLINICAL TRIAL: NCT04720079
Title: The Effectiveness of Thoracic Paravertebral Block in Improving the Anesthetic Effects of Regional Anesthesia for Upper Extremity Arteriovenous Fistula Surgery
Brief Title: Paravertebral Block With Brachial Plexus Block for Upper Arm Arteriovenous Fistula Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2303
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2021-11

CONDITIONS: Regional Anesthesia Success

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostobrachial nerve Infiltration (Active Comparator): Preoperative infiltration of intercostobrachial nerve with 10ml of ropivacaine 0.5%
  Interventions: Procedure: Subcutaneous infiltration of intercostobrachial nerve
- Ultrasound guided T2 paravertebral block (Active Comparator): Preoperative ultrasound guided T2 paravertebral nerve block with 10ml of ropivacaine 0.5%
  Interventions: Procedure: T2 paravertebral nerve block

INTERVENTIONS:
Procedure: Subcutaneous infiltration of intercostobrachial nerve — Preoperative subcutaneous infiltration of intercostobrachial nerve with 10ml of 0.5% ropivacaine
  Arms: Intercostobrachial nerve Infiltration
Procedure: T2 paravertebral nerve block — Preoperative ultrasound guided T2 paravertebral nerve block with 10ml of 0.5% ropivacaine
  Arms: Ultrasound guided T2 paravertebral block

SUMMARY:
The primary goal of this quality improvement project is to find the optimal surgical conditions for patients undergoing upper arm arteriovenous graft surgery. Currently, there are two anesthetic techniques used in clinical practice. The goal is to standardize future practice and improve the care of patients postoperatively. The two techniques used in conjunction with a brachial plexus block are paravertebral nerve block and subcutaneous infiltration.

DETAILED DESCRIPTION:
This study is designed to test the null hypothesis that paravertebral nerve block or subcutaneous infiltration provide similar operating conditions when combined with supraclavicular nerve block for upper arm arteriovenous fistula surgery. The results will help determine which approach to use and guide future research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) undergoing upper limb arteriovenous fistula surgery at UNC Chapel Hill hospital

Exclusion Criteria:

* Contraindication to regional anesthesia
* Significant peripheral neuropathy or neurological disorder of the upper extremity
* Cognitive or psychiatric condition that will interfere with patient assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Successful Regional Anesthesia | By end of surgery
  Success is considered a regional anesthetic without rescue analgesic medications (including surgeon administered local anesthetic) or conversion to general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grant, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC